CLINICAL TRIAL: NCT05753813
Title: Exploring the Effects of an Intravaginal Lactic Acid Gel on the Vaginal Microbiome
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Queen's Medical Center (Other)
Collaborators: University of Hawaii Foundation (Unknown)
Responsible Party: Principal Investigator, Olivia Manayan, MD MPH, PGY-2, University of Hawaii Ob/Gyn Residency, Queen's Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RA-2022-015
Record Dates: First submitted 2023-01-04; First posted 2023-03-03 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Bacterial Vaginosis; Vulvovaginal Candidiasis
MeSH Terms: conditions — Vaginosis, Bacterial; Candidiasis, Vulvovaginal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Study group (Experimental): This is a single-arm study. all participants are assigned to this arm. all study participants will receive Phexxi, the study drug. 8 pre-filled vaginal inserters with vaginal gel, Phexxi, will be provided to each of the participants with verbal and written instructions for application. Patients will be instructed to use Phexxi twice per week, on the same days every week.
  Interventions: Drug: Phexxi

INTERVENTIONS:
Drug: Phexxi — intravaginal gel twice weekly for 4 weeks.

SUMMARY:
This project aims to investigate if the contraceptive method, Phexxi, causes changes to the composition of the vaginal microbiome. The investigators hypothesize that regular use of Phexxi will cause increased colonization of lactic acid-producing lactobacilli, which could have positive effects in the way of preventing recurrent episodes of BV and candida infections.

DETAILED DESCRIPTION:
This is a single center, prospective trial, which comprises of a pre-post study design that will be looking at the vaginal microbiome makeup of participants before and after a four-week course of Phexxi. The primary outcomes will be an increase in lactic acid-forming lactobacilli, as well as a decrease in patient-reported symptoms of vulvovaginitis.

This study will be based at the Queen's Medical Center (QMC), POB1 Suite 1004. Eligible patients will be approached by participating clinicians (all doctors providing care at the 1004 clinic) to assess interest in study participation.. The principal investigator will review the weekly schedule for the 1004 clinic and alert the attending physicians of patients who may be eligible for the study based on chart review. A HIPAA waiver will be required for this stage of recruitment, as the principal investigator would otherwise not be accessing these patient's charts. The attending physician staffing the 1004 clinic will ask the flagged patients if they are interested in learning about the study and review general study objectives with patients. If the patient is interested in participating, the research associates will approach the patient to more thoroughly screen, then conduct the informed consent process. Informed consent will be collected from every participant prior to the start of the study.

After obtaining informed consent, the research team will review standardized instructions for using the study medication with the patient and the research associate will provide a take-home kit including all of the study materials, including instructions for collecting each swab and for returning the samples. Samples will be self-collected by participants at their home at intervals specified in the study instructions. All materials provided to the patient will be pre-labeled with their study ID, protecting each participant's PHI. No collections will take place in-clinic. These materials include all surveys, patient's diary, and all swab vials. The three collection points are as follows: 1) baseline, prior to starting intervention (see below for recommendations on collecting baseline swab), 2) after completion of the intervention (30 days after baseline collection), and 3) 30 days after completion of the intervention (60 days after baseline collection).

All vaginal swabs must be frozen within 48 hours of collection. As such, the participants will be asked to send their samples within 24 hours in order to give adequate time for delivery to the storage facility and be asked to collect their specimens between Sunday and Thursday so samples can reach the facility during business hours. Freezing will occur at the research site. Each patient's study kit will include a prepaid shipping envelope, which the participant can use to mail or drive their specimen to the research team who will then place it in the freezer until it is ready for analysis.

The first phase of the study will include an assessment and classification of patients' vaginal microbiome prior to receipt of the intervention. To get the best representation of the participant's baseline microbiome, the participant will be asked to collect their baseline swab no sooner than 10 days after menses, as menses-induced changes in the microbiome have been shown to resolve after this time12. For similar reasons, if participants are being treated with an acute course of antibiotics or antifungals at the time of recruitment, they will be asked to wait 10 days after the completion of their medication course before collecting their baseline swab. There will be two additional time points for collection: collection 2) at the end of the 30 day intervention, and collection 3) 30 days after completion of the intervention.

Once received at the research site, samples will be stored in a specimen freezer at -80 degrees F until all specimens are received, at which point they will analyzed using NextGen sequencing, a DNA sequencing technology that will identify the genetic makeup of their specimens. This will be done to sequence the genome of the bacteria of the microbiome, not the patient's genetic material. The first phase of the study will also include a survey, which will collect demographic information from each participant, as well as assess patients' current acceptability of a vaginal gel for prophylactic use, their most bothersome symptoms, and how their quality of life is affected by recurrent vulvovaginitis. The specific information collected from each participant can be found below in Data Analysis. The survey used to measure this will be the Vulvovaginal Symptom Questionnaire (VSQ), which has been validated for the purposes stated above. There will also be an added space in the survey provided for open-ended answers and comments.

Measurement for primary outcomes will be done using two separate methods. In order to assess for the presence of lactic acid-forming organisms before and after the lactic acid gel intervention, NextGen DNA sequencing will be completed on self-collected samples submitted by participants. The analysis of these samples will be performed by Dr. Miller, at an in-house lab run by the UH Maternal Fetal Medicine division. In order to assess for patient-experienced symptoms, survey B will be administered prior to, immediately after, and 30 days after intervention.

In order to measure our secondary outcome, Survey C will be administered at collection points 2 and 3 of the vaginal swabs. This survey is a validated tool to assess for the acceptability, appropriateness, and feasability of an intervention (Acceptability of Intervention Measure, or AIM, Intervention Appropriateness measure, or IAM, and Feasibility of Intervention Measure, or FIM).

The intervention will take place on a rolling basis, as patient participation will have no bearing on other participants. The intervention itself will take place over thirty days. 8 pre-filled vaginal inserters with vaginal gel, will be provided to each of the participants with verbal and written instructions for application. Patients will be instructed to use Phexxi twice per week, on the same days every week. Throughout the 30 days, participants will also be asked to keep a diary of events occurring when they used the product, such as intercourse or menses, as well as record any symptoms or side effects they noticed when using the product. The diary can be sent back with the second specimen vial. Disposal of the product may be done in a regular waste basket.

Approximately 30 days after completion of the intervention, participants will receive an email reminder to collect and send a third collection swab in for analysis. This email will also include the link for the third and final set of surveys.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-54
* Female
* Pre-menopausal
* Can speak and read in English
* Displays capacity for informed consent
* Has had 2 or more documented and/or self-reported episodes of symptomatic BV or candida infection in the last year, requiring, over-the-counter or prescription treatment

Exclusion Criteria:

* Pregnant or trying to become pregnant
* Post-menopausal
* Using NuvaRing device
* A past medical history of kidney disease, recurrent UTI, and/or urinary tract abnormalities
* Current UTI
* Using Phexxi as a contraceptive during the collection period of the study

Ages: 18 Years to 54 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
To assess participant's baseline vaginal microbiome makeup | Within one week of recruitment, unless menstruating. If this is the case, the participant will be asked to wait 10 days from the cessation of menses in order to allow restoration of baseline vaginal microbiome
  NextGen analysis pre-intervention
To assess if the use of Phexxi causes changes in the vaginal microbiome from baseline after thirty days of use | 30 days after baseline vaginal swab collection
  NextGen analysis immediately post-intervention
To assess if the use of Phexxi causes changes in the vaginal microbiome | 60 days after baseline vaginal swab collection
  NextGen analysis 30 days post-completion of intervention
To assess participant's baseline vulvovaginitis symptoms | On day of recruitment to the study
  Survey to be completed pre-intervention
To assess if the use of Phexxi decreases vulvovaginitis symptoms in study participants | 30 days after baseline vaginal swab collection
  Survey to be completed immediately post-intervention. This survey is a validated tool to assess for symptoms of vulvovaginitis (Vulvovaginal Symptoms Questionnaire, or VSQ). It employs a binary scoring system, giving 0 points for no and 1 point for yes, with 21 questions which assess vulvovaginitis symptoms.
To assess if the use of Phexxi decreases vulvovaginitis symptoms in study participants | 60 days after baseline vaginal swab collection
  Survey to be completed 30 days post-completion of intervention. This survey is a validated tool to assess for symptoms of vulvovaginitis (Vulvovaginal Symptoms Questionnaire, or VSQ). It employs a binary scoring system, giving 0 points for no and 1 point for yes, with 21 questions which assess vulvovaginitis symptoms.

SECONDARY OUTCOMES:
To assess patient satisfaction/acceptability of this intervention as a therapeutic/prophylactic agent for recurrent vulvovaginitis | 30 and 60 days after baseline swab collection
  Survey at 2 time points: immediately post-intervention, and 30 days post-completion of intervention. This survey is a validated tool to assess for the acceptability, appropriateness, and feasability of an intervention (Acceptability of Intervention Measure, or AIM, Intervention Appropriateness measure, or IAM, and Feasibility of Intervention Measure, or FIM). It lists a number of statements to assess the above measures and asks the participant to circle the ones which apply to them.

CONTACTS AND LOCATIONS:
Overall Officials: Olivia Manayan, MD, MPH, Principal Investigator — University of Hawaii; Bliss Kaneshiro, MD, MPH, Principal Investigator — Queen's Medical Center; Corrie Miller, DO, Principal Investigator — University of Hawaii
Locations (1):
- Queens Medical Center, 1004 Clinic POB1, Honolulu, Hawaii, United States

IPD SHARING:
Plan to Share IPD: No
Patient information will be de-identified and connected to a unique Study ID. All identifiable information will be stored in a password protected and encrypted computer in the PI's research office at QMC, which is secured at the 1004 clinic. The signed consent forms will also be stored at the 1004 clinic, in a folder located in a locked office. Only the PI and Dr. Kaneshiro will have access to the identifiable information. Dr. Miller, who will be performing analysis using specimens prelabeled with the study ID, will not have access to participant PHI.
  If participants opt, in their initial consent, to receive a copy of their vaginal microbiome results, the results will be sent to them via email, using a QMC email address. In order to encrypt this email, the function [encrypted] will be placed in the subject line.

DOCUMENTS (2):
  • Study Protocol (2022-11-23): https://cdn.clinicaltrials.gov/large-docs/13/NCT05753813/Prot_000.pdf
  • Informed Consent Form (2022-12-12): https://cdn.clinicaltrials.gov/large-docs/13/NCT05753813/ICF_001.pdf